CLINICAL TRIAL: NCT02889770
Title: Dead Space Monitoring During PEEP Titration in Patients With Hypoxemia Secondary to Acute Respiratory Distress Syndrome
Brief Title: Dead Space Monitoring With Volumetric Capnography in ARDS Patients
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Emiliano Gogniat, Physical therapist, Hospital Italiano de Buenos Aires
Other Study IDs: 1968
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Acute Respiratory Distress Syndrome; Capnography
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: PEEP titration — Exposure to different PEEP levels

SUMMARY:
This studies´ objective is to describe how different PEEP levels affect dead space measured by Bohr´s formula.

DETAILED DESCRIPTION:
In ARDS patients PEEP has contradictory effects on ∆P (driving pressure of the airway) hat depends on the balance between lung recruitment and overdistension. Some authors showed that incremental levels of PEEP did not much affect dead space in ARDS patients. These studies used different methods for the assessment of dead space.

Such technique also overestimates the dead space. We believe that the right way to measure dead space is applying the original Bohr's equation using the mean PACO2 value. Therefore, the aim of this observational study was to describe the effect that PEEP has on Bohr's dead space and its sub-components in mechanically ventilated patients with ARDS.

This observational study was performed in the Intensive Care Unit of a University Hospital.

Protocol design The protocol started recording the data during baseline protective ventilation. After 15 minutes of data recording, we studied four levels of PEEP - 0, 6, 10 and 16 cmH2O - which were randomly assigned by a randomization table.

Respiratory, hemodynamic, arterial blood gas analysis and volumetric capnographic parameters were recorded. We analyzed the last 2 minutes of each protocol steps consisting in more than 30 breaths or data-points.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* requirement of invasive mechanical ventilation for more than 4 hours and less than 12 hours
* severe hypoxemia (PAFI < 200) secondary to ARDS or post-operatory atelectasis

Exclusion Criteria:

-requirement of invasive mechanical ventilation prior to enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Dead space variation | 60 min
  How dead space, measured by Bohr´s formula, varies with different PEEP levels during a recruitment manouver

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Gogniat, PT, Principal Investigator — Hospital Italiano de Buenos Aires

IPD SHARING:
Plan to Share IPD: Undecided